CLINICAL TRIAL: NCT07331948
Title: INFLUENCE OF VOJTA THERAPY ON POSTURAL CONTROL AND MANIPULATION IN CEREBRAL PALSY INFANTILE HEMIPARESIS
Brief Title: INFLUENCE OF VOJTA THERAPY IN CEREBRAL PALSY. INFANTILE HEMIPARESIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Integral Kaplan (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0207202326323
Record Dates: First submitted 2025-12-27; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Pediatric Hemiparesis
Keywords: Hemiparesis, Pediatric hemiparesis, Vojta therapy , Physiotherapy, Pediatric rehabilitation, Upper limb function, Box and Block Test, EEG, EMG
MeSH Terms: conditions — Paresis

STUDY DESIGN:
Intervention Model Description: Single-case, single-group interventional study in which one pediatric participant with hemiparesis receives a Vojta therapy session and outcomes are measured before and after the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vojta Therapy (Experimental): One intensive physiotherapy session based on the Vojta method, delivered by a physiotherapist specialized in Vojta therapy in an outpatient clinic
  Interventions: Other: Vojta therapy session

INTERVENTIONS:
Other: Vojta therapy session — One intensive physiotherapy session based on the Vojta method, including standardized reflex locomotion stimulation patterns, delivered by a physiotherapist specialized in Vojta therapy in an outpatient clinic

SUMMARY:
This study describes a single pediatric case with hemiparesis who received a specialized physiotherapy intervention based on the Vojta method. The child, aged 15 years, was treated in a clinical setting by a physiotherapist certified in Vojta therapy during one intensive treatment session. Upper limb function was evaluated before and after the intervention using the Box and Block Test, as well as electroencephalography (EEG) and electromyography (EMG) recordings to explore changes in motor control and brain activity. The main purpose of this study is to document the feasibility and short-term effects of a Vojta-based physiotherapy session on upper limb function and neurophysiological parameters in a child with hemiparesis

DETAILED DESCRIPTION:
This single-case clinical study involves a 15-year-old child with hemiparesis who underwent a physiotherapy intervention using the Vojta method in an outpatient clinic. The intervention consisted of one intensive treatment session delivered by an experienced physiotherapist specialized in Vojta therapy, following standardized stimulation patterns tailored to the patient's motor profile. Upper limb function was assessed immediately before and after the intervention using the Box and Block Test, while simultaneous EEG and EMG recordings were obtained to characterize cortical and muscular activation during motor tasks. The primary objective is to evaluate short-term changes in manual function, and the secondary objective is to describe associated neurophysiological changes, to generate hypotheses for future clinical trials in pediatric patients with hemiparesis.

ELIGIBILITY:
Inclusion Criteria:

* Hemiparesis, 0-16 years, cognitive ability to perform the Box and Block Test

Exclusion Criteria:

* Severe musculoskeletal deformities or pain in the upper limb that prevent the performance of the Box and Block Test, Severe visual or auditory impairment that prevents understanding or performing the Box and Block Test

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2024-01-22 (Actual); Primary Completion 2024-01-22 (Actual); Study Completion 2024-01-22 (Actual)

PRIMARY OUTCOMES:
Change in upper limb manual dexterity (Box and Block Test) | Baseline and immediately after the Vojta therapy session
  Manual dexterity of the affected upper limb will be assessed using the Box and Block Test. Higher scores indicate better manual dexterity

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Kaplan, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because this is a single-case study and the data are potentially identifiable, making it difficult to fully protect the participant's privacy.

REFERENCES:
- [Background] Sanz-Esteban I, Calvo-Lobo C, Rios-Lago M, Alvarez-Linera J, Munoz-Garcia D, Rodriguez-Sanz D. Mapping the human brain during a specific Vojta's tactile input: the ipsilateral putamen's role. Medicine (Baltimore). 2018 Mar;97(13):e0253. doi: 10.1097/MD.0000000000010253. PMID 29595683
- See also: Related Info — https://www.centrokaplan.es